CLINICAL TRIAL: NCT05311111
Title: Efficacy and Safety of the Distal Radial Approach in Percutaneous Coronary Interventions: Protocol of a Randomized Controlled Non-inferiority Trial
Brief Title: Efficacy and Safety of the Distal Radial Approach
Acronym: TunDRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Administration of Military Health, Tunisia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: santemilitaire7
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Vascular Access Complication; Coronary Artery Disease
Keywords: Radial artery; coronary angiography; percutaneous coronary intervention; safety; efficacy; radial approach; anatomical snuff box
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-blind, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: single blind during the analyze
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- distal radial artery approach (Experimental): Elective percutaneous coronary intervention by forearm radial artery through the distal radial artery in the dorsum of the hand or the anatomical snuff-box
  Interventions: Procedure: distal radial artery approach
- conventional radial artery approach (Active Comparator): Elective percutaneous coronary intervention through conventional radial artery access
  Interventions: Procedure: conventional radial artery approach

INTERVENTIONS:
Procedure: distal radial artery approach — Procedure: Use of radial artery for access for a coronary angiography or intervention After preparation and local anesthesia, the operator will puncture the distal radial artery in the dorsum of the hand or the anatomical snuff-box. Then a sheath will be placed. A cocktail combining Risordan®, Loxen® and unfractionated heparin will be injected through the sheath. a wire will be introduced. At the end of the procedure, the sheath will be removed immediately and hemostasis by compression will be carried out with an elastic band for 12 hours. The choice of limb side, sheath, catheters will be chosen according to the operator's discretion.
  Other Names: DRA
  Arms: distal radial artery approach
Procedure: conventional radial artery approach — Procedure: conventional radial access for a percutaneous coronary intervention After preparation and local anesthesia, the operator will puncture the proximal radial artery at the conventional site in distal forearm. Then a sheath will be placed. A cocktail combining Risordan®, Loxen® and unfractionated heparin will be injected through the sheath. a wire will be introduced. At the end of the procedure, the sheath will be removed immediately and hemostasis by compression will be carried out with an elastic band for 12 hours. The choice of limb side, sheath, catheters will be chosen according to the operator's discretion.
  Other Names: TRA
  Arms: conventional radial artery approach

SUMMARY:
The aim of this non-inferiority trial is to determine if the distal radial access (DRA) during percutaneous coronary intervention (PCI) has an acceptable efficacy compared to the reference access through the conventional radial artery (TRA) with a lower rate of radial artery occlusion (RAO) in real life practice.

DETAILED DESCRIPTION:
The conventional radial approach is the recommended vascular access for percutaneous coronary interventions. It is effective, feasible, but associated with a risk of occlusion of the radial artery.

The distal radial approach is proposed as a new approach to reduce complications and preserve the radial artery. However, few clinical trials in real life were conducted in North African patients.

This trial aims to evaluate the efficacy and safety of the distal radial approach versus the conventional radial approach.

This trial is a non-inferiority, randomized controlled trial with two parallel arms: distal radial approach and conventional radial approach. Two hundred and fifty patients scheduled for percutaneous coronary intervention will be included. The two main endpoints are the puncture success rate with a non-inferiority margin of 10% and the rate of 30-day occlusion of the punctured radial artery.

Secondary endpoints: catheterization success, crossover rate, procedure time, radial artery spasm, bleeding complications, QuickDASH score, pain score and operator satisfaction A single blind analysis will be led according to the per-protocol and intention-to-treat methods.

Avoiding occlusion of the puncture site allows to preserve the radial artery for subsequent coronary or cerebral percutaneous interventions as well as for coronary bypasses and hemodialysis fistulas. The results will provide the parameters related to the efficacy and safety of the distal radial approach, so improving clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Hospitalized in the cardiology department of the military hospital of Tunis.
* elective Percutaneous coronary intervention performed by experienced operators or fellows trained in the proximal and distal radial approach

Non-inclusion criteria:

* not provided written informed consent
* both radial arteries were used for prior catheterization
* Under oral anticoagulation
* Having coronary bypass surgery
* Hemodynamic instability
* contra-indication to the radial approach:

  * Orthopedic surgery: amputation
  * Severe burns of both upper limbs.
  * Radial artery pulse not palpable, negative modified Allen test or Barbeau classification type D
  * Identified radial vascular anomaly: stenosis, fistula, tortuosity not allowing passage of the catheter

Exclusion Criteria:

* death within a short period of time after admission
* PCI by the same puncture site will be performed within 30 days after the first puncture
* lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Puncture success rate | During the procedure
  Comparison of Puncture success rate between two groups: Distal Radial Access (DRA) and conventional Trans Radial Access (TRA)
Radial artery occlusion rate | 30 days
  Use of ALLEN and Barbeau tests, if abnormal, color Doppler ultrasound to assess the patency of the radial artery will be realized.

SECONDARY OUTCOMES:
Crossover rate | During the procedure
  Comparison of the access site crossover rate in each group to complete the staged procedure
Duration of the puncture | During the procedure
  Exact measurement of puncture duration in seconds
Radial artery spasm | During the procedure
  The incidence of vasospasm that necessitates additional medication or forces access site cross over is registered
Number of patients presenting hematoma | 24 hours
  Hematoma according to Early Discharge After Transradial Stenting of Coronary Arteries Study (EASY) score, The score ranges from 1 (≤5 cm diameter) to 5 ( ischemic threat of the hand).
Pain scale | 24 hours
  through 0-10 numeric pain rating scale, 0 being no pain and 10 being the worst pain imaginable
QuickDASH questionnaire | 30 days
  The Quick-Disabilities of the Arm, Shoulder and Hand (QuickDASH) score is used to assess hand function. The score ranges from 0 (no disability) to 100 (most severe disability)
Operator satisfaction | at the end of the inclusion
  through 0-10 rating scale; 0 being very dissatisfied; 0 being very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Aymen Noamen, MD, Principal Investigator — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis; Nadhem Hajlaoui, Pr, Study Director — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis; Wafa Fehri, Pr, Study Chair — military hospital of Tunis , Tunis EL manar University, Faculty of medicine of Tunis
Locations (1):
- Military hospital of Tunis, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben Amara A, Noamen A, Anouar Y, Chenik S, Hajlaoui N, Fehri W. Evaluation of the Distal Radial Approach in percutaneous coronary interventions. Controlled, randomized non-inferiority trial. Tunis Med. 2022 mars;100(3):192-202. PMID 36005910